CLINICAL TRIAL: NCT02244437
Title: Ibuprofen vs Acetaminophen in the Prevention of Acute Mountain Sickness: A Double Blind, Randomized Controlled Trial
Brief Title: Ibuprofen vs Acetaminophen for AMS Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mountain Medicine Society of Nepal (Other)
Responsible Party: Principal Investigator, Buddha Basnyat, Dr, Mountain Medicine Society of Nepal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202/2013
Record Dates: First submitted 2014-09-14; First posted 2014-09-19 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Acute Mountain Sickness, Blood Oxygen Saturation, Headache
Keywords: altitude, altitude illnesses, headache
MeSH Terms: conditions — Altitude Sickness; Headache | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibuprofen (Active Comparator): Ibuprofen has been shown to prevent AMS from previous studies.
  Interventions: Drug: Ibuprofen
- Acetaminophen (Experimental): Acetaminophen has not been tested yet in AMS prevention.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen
  Other Names: 600 mg per oral three times in a day
  Arms: Ibuprofen
Drug: Acetaminophen
  Other Names: 1g per oral three times in a day
  Arms: Acetaminophen

SUMMARY:
AMS (acute mountain sickness) affects those who ascend too high (>2000m) too fast. Acetazolamide is an effective drug for the prevention of AMS where proper acclimatization with gradual ascent may not be an option. AMS presents with headache and other non-specific symptoms such as nausea, tiredness, and dizziness. Because of the side effects of acetazolamide such as a tingling sensation, other drugs have been investigated to see if they will prevent AMS. Ibuprofen has recently been shown to prevent AMS. In this present study the investigators want to see if acetaminophen can also prevent AMS as acetaminophen unlike ibuprofen does not have gastric side effects. Second, because acetaminophen has much less anti-inflammatory component than ibuprofen, it may also provide some insight into the pathophysiology of AMS if acetaminophen were found to be effective in the prevention of AMS.

DETAILED DESCRIPTION:
Acute mountain sickness (AMS) is a well-known disorder in sojourners to high altitude (>2000m) characterized by headache, nausea and tiredness, akin to hangover-like symptoms. The Lake Louise criteria for AMS was primarily developed to allow uniformity in comparing the prevalence of AMS in different high altitude regions.

Proper acclimatization by gradual ascent to high altitude is the best means of prevention of AMS. However there may be instances when rapid ascents may be necessary. Acetazolamide is the best known drug for the prevention of AMS. Because of its well-known side effects like tingling sensation in the fingers and toes and its potential sulpha allergy (acetazolamide is a sulpha-based drug) problems, alternative drugs in the prevention of AMS have been sought. Recently two randomized controlled trials have shown the usefulness of ibuprofen 600 mg tid orally in the prevention of AMS.

The exact mechanism causing AMS is unknown although evidence points to a process in the central nervous system. The mechanism of headache, the main feature in most AMS patients, is probably multifactorial with various chemical and mechanical factors activating a final common pathway, the trigeminovascular system. Triggering factors associated with high altitude hypoxia leading to AMS may include arachidonic acid metabolites amongst others such as serotonin, histamine, and nitric oxide. The response in AMS prevention to non-steroidal anti-inflammatory drugs (NSAIDs) and steroids provides indirect evidence of arachidonic acid pathway and inflammation in the genesis of AMS.

But in contrast, the role of drugs such as acetaminophen which primarily provide analgesia by blunting the meningovascular receptors known to mediate nociception is unknown in the prevention of AMS. Crucially if acetaminophen can prevent AMS the gastric irritation and possible gastrointestinal bleeding which are well known side effects of ibuprofen would not be encountered. In addition acetaminophen like ibuprofen and (unlike acetazolamide) is easily available over the counter.

Therefore, the investigators hypothesize that acetaminophen in adequate dosage ( 1 g tid) will be as effective as ibuprofen ( 600 mg tid) in the prevention of AMS.

Western trekkers will be randomly administered either acetaminophen or ibuprofen in a double blind fashion at 4300m where the investigators will enroll the participants. Then, at 5000 m at Lobuje after 48 to 96 hours the investigators will re-examine with the Lake Louise Questionnaire (LLQ) to see their AMS status. The investigators will also check the pulse oximeter.

Sample Size:

With a variable alpha 5%, power 80%, control 34% (based on previous studies) and experimental group 18%, the sample size arrived at (using http://www.sealedenvelope.com/power/binary-superiority/ ) was 115 per arm, a total of 230 participants. With a 20 % drop out the final number the investigators require is 288 participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between the ages of 18 and 65, male or female, non-Nepali, without AMS or any concurrent illness, and not already taking NSAIDs and acetazolamide or any other drug for the prevention of altitude illness. Subjects will be enrolled by study administrators en route directly to Everest Base Camp or Kala Patthar between the villages of Pheriche/Dingboche and Lobuche.

Exclusion Criteria:

* Individuals not meeting inclusion criteria, including mild AMS (more than one mild symptom on the Lake Louise Questionnaire) or significantly depressed oxygen saturation (<75%); females known to be pregnant, cannot exclude the possibility of being pregnant, or have missed menses by over 7 days; individuals who have spent 24 hours at an altitude of 4500 meters/14,000 feet within the last 9 days; anyone known to have taken any of the following in the last 2 days: acetazolamide (Diamox®), steroids (dexamethasone, prednisone), theophylline, or diuretics (Lasix®); individuals who have a known intracranial space occupying lesion or a history of elevated intracranial pressure, (i.e. tumors, hydrocephalus, etc).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Acute Mountain Sickness (AMS) | Upon reaching 5000m altitude (Lobuche) of Nepal Himalaya. Average stay of the trekkers at this altitude is expected about a day or more. The assessment of the participants will be done next day (after spending overnight) upon their arrival.
  AMS diagnosis will be done using Lake Louise Questionnaire (LLQ) which requires a score of three or greater with the mandatory presence of headache and at least one of the following symptoms: dizziness or light-headedness, fatigue, gastrointestinal (GI) symptoms (nausea/vomiting), or difficulty sleeping.
  LLQ is a self-report symptom questionnaire and it will be assessed among all the study participants upon arrival to the study end point i.e. 5000m altitude (Lobuche) as specified above.

SECONDARY OUTCOMES:
Blood Oxygen Saturation (SPO2) | Upon reaching 5000m altitude (Lobuche) of Nepal Himalaya. Average stay of the trekkers at this altitude is expected about a day or more. The assessment of the participants will be done next day (after spending overnight) upon their arrival.
  Blood oxygen saturation (percentage of oxygen in the blood) among all the study participants will be measured using Pulse Oximetry. The percentage of oxygen in the blood measured will be abbreviated as SPO2 in the spreadsheet.
Heart Rate (HR) | Upon reaching 5000m altitude (Lobuche) of Nepal Himalaya. Average stay of the trekkers at this altitude is expected about a day or more. The assessment of the participants will be done next day (after spending overnight) upon their arrival.
  Heart rate (HR) will be assessed among all the study participants using Pulse Oximetry. The heart rate measured in the study will be abbreviated as HR in the spreadsheet.
High Altitude Headache (HAH) | Upon reaching 5000m altitude (Lobuche) of Nepal Himalaya. Average stay of the trekkers at this altitude is expected about a day or more. The assessment of the participants will be done next day (after spending overnight) upon their arrival.
  High altitude headache (HAH) and its severity will be scored based on a Visual Analog Scale (VAS) and the headache score identified on the designated LLQ score upon arrival to the study end point i.e. 5000m altitude (Lobuche).

CONTACTS AND LOCATIONS:
Overall Officials: Buddha Basnyat, MD, Principal Investigator — Mountain Medicine Society of Nepal (MMSN), Nepal International Clinic (NIC) and Oxford University Clinical Research Unit (OUCRU), Kathmandu, Nepal; Matiram Pun, MBBS/MSc/MA, Principal Investigator — Mountain Medicine Society of Nepal (MMSN) and Department of Clinical Physiology, Maharajgunj Medical Campus, Institute of Medicine (IOM), Kathmandu, Nepal; Nicholas C Kanaan, MD, Principal Investigator — Department of Surgery, Division of Emergency Medicine, University of Utah, Salt Lake City, UT, USA
Locations (1):
- Buddha Basnyat, MD, Kathmandu, Nepal